CLINICAL TRIAL: NCT04114825
Title: A Phase 2, Double-Blind, Placebo Controlled Study of RV001V in Men With Biochemical Failure Following Curatively Intended Therapy For Localized Prostate Cancer (BRaVac)
Brief Title: Study of RV001V in Biochemical Failure Following Curatively Intended Therapy For Localized Prostate Cancer
Acronym: BRaVac
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RhoVac APS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RhoVac-002
Record Dates: First submitted 2019-09-28; First posted 2019-10-03 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer Recurrent
Keywords: Biochemical relapse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RV001V (Experimental): Total of 12 SC vaccinations with RV001V. The first 6 vaccinations (priming period) will be given every 2 weeks, and then the following 5 vaccinations (7 through 11) will be administered with 4 weeks between each vaccination (Maintenance period), and the last vaccination (12th) will be administered 6 months following the 11th vaccination (boosting injection).
  Interventions: Biological: RV001V
- Placebo (Placebo Comparator): Total of 12 SC vaccinations with placebo. The first 6 vaccinations (priming period) will be given every 2 weeks, and then the following 5 vaccinations (7 through 11) will be administered with 4 weeks between each vaccination (Maintenance period), and the last vaccination (12th) will be administered 6 months following the 11th vaccination (boosting injection).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: RV001V — RV001V consists of the peptide RV001 and the adjuvant Montanide ISA 51. RV001 Vaccine 0.1 mg/mL (RV001V).
  Arms: RV001V
Other: Placebo — Placebo consist of the vaccine vehicle and the adjuvant Montanide ISA 51. Placebo
  Arms: Placebo

SUMMARY:
This Phase II trial will enroll approximately 180 adult male patients with an earlier histologic diagnosis of prostatic adenocarcinoma and a biochemical recurrence (BCR) within 3 years of radical prostatectomy (RP) or definitive RT and no distant metastasis or locoregional recurrence. The trial is a randomized placebo-controlled double-blind study of a peptide cancer vaccine (RV001V).

ELIGIBILITY:
Main Inclusion Criteria:

* Biochemical recurrence (BCR) within 3 years of radical prostatectomy (RP) or definitive RT and no distant metastasis by standard CT imaging and bone scintigraphy, or locoregional recurrence (including lymph nodes) assessed by CT or multi-parametric magnetic resonance imaging (MRI) and confirmed with negative biopsy in case of prior RT.
* In case of BCR after RP all the following criteria should apply: a. PSA ≥0.2 ng/mL, b. PSA Doubling Time (PSADT) >3 months and <12 months
* In case of BCR after RT all the following criteria should apply: a. PSA >nadir + 2 ng/mL, b. PSADT >3 months and <12 months
* ECOG performance status ≤2.
* Laboratory values obtained ≤30 days prior to first vaccination: Hemoglobin ≥5.6 mmol/L; Absolute granulocyte count ≥1.5 x 109 /L, Platelets ≥100 x 109 /L., Total bilirubin ≤1.5 x upper limit of normal (ULN).
* Creatinine ≤1.5 x ULN.
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤2.5 x ULN.

Main Exclusion Criteria:

* Patients who are receiving androgen-deprivation therapy or considered a candidate for immediate anti-androgen deprivation therapy (ADT) as judged by the investigator.
* Patients who have received prior ADT are not eligible with the exception of those that received ADT ≤36 months in duration and ≥9 months before randomization and administered only in the neoadjuvant/adjuvant setting.
* Patient is planned for salvage therapy with RT or radical prostatectomy.
* Castrate level of serum testosterone <50 ng/dL at screening.
* PSA >10 ng/mL

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Time to PSA progression | Up to 3 years
  Time to PSA progression is defined as the time from randomization to doubling of PSA from the baseline value. The time to doubling will be estimated from a log-linear regression of PSA values.

SECONDARY OUTCOMES:
Safety by frequency and severity of adverse events (AEs) | Up to 16 months
  The numbers and proportions of patients with any treatment-emergent adverse event (TEAE), and any serious TEAE will be summarized
Time to initiation of a subsequent antineoplastic therapy | Up to 3 years
Proportion of patients showing a PSA response from baseline | Up to 3 years
Disease-free survival (DFS) | Up to 3 years
  time from randomization to documented clinical recurrence (distant or local), or death from any cause, censoring at date of last follow-up (FU)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Brasso, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (36):
- United States (7):
  - Tampa Bay Medical Research, Clearwater, Florida
  - Chesapeake Urology Research Associates, Towson, Maryland
  - GU Research Network/Urology Cancer Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Icahn School of Medicine at Mount Sinai Hospitals, New York, New York
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - The Urology Place, San Antonio, Texas
- Belgium (3):
  - Gent University Hospital, Ghent
  - CHU de Liège, Liège
  - Hôpital Erasme, Liège
- Denmark (6):
  - Aalborg University, Departmen of Urology, Aalborg
  - Aarhus University Hospital, Department of Urology, Aarhus
  - Rigshospitalet, Copenhagen Prostate Cancer Center, Copenhagen
  - Herlev & Gentofte Hospital, Department of Urology, Herlev
  - Urinvejskirurgisk afdeling, Hospitalsenheden Vest, Holstebro
  - Odense University Hospital, Deparment of Urology, Odense
- Finland (5):
  - Meilahti Tower Hospital, Helsinki
  - Oulu University Hospital, Oulu
  - Seinajoki Central Hospital, Seinäjoki
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku
- Germany (6):
  - University Hospital Dresden, Dresden
  - Urologicum Duisburg, Duisburg
  - Urologische Praxis Dr. Wolfgang Warnack, Hagenow
  - Urologische Praxis. M. Markov, Halle
  - Studienpraxis Urologie, Nürtingen
  - University Hospital Tuebingen, Tübingen
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Skåne University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Umeå University Hospital, Umeå
- United Kingdom (4):
  - Clatterbridge Centre for Oncology, Liverpool
  - Royal Free London NHS Foundation Trust Royal Free Hospital, London
  - Nottingham University Hospital, Nottingham
  - University Hospital Southampton, Southampton